CLINICAL TRIAL: NCT06431282
Title: In Vivo Visualisation of Hyaluronic Acid After CO2 Laser Compared to Thulium Laser Treatment
Brief Title: Hyaluronic Acid Delivery: CO2 Laser Versus Thulium Laser Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Lynhda Nguyen, Principle Investigator, Universitätsklinikum Hamburg-Eppendorf
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 01-24
Record Dates: First submitted 2024-02-19; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Aging Skin
MeSH Terms: interventions — Lasers, Gas

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CO2 laser + HA (Active Comparator): Probands are treated with a CO2 laser. Afterwards a HA gel will be applied.
  Interventions: Other: CO2 laser + HA
- Thulium laser + HA (Active Comparator): Probands are treated with a thulium laser. Afterwards a HA gel will be applied.
  Interventions: Other: Thulium laser + HA

INTERVENTIONS:
Other: CO2 laser + HA — Probands will be treated with a CO2 laser. Afterwards a HA gel will be applied. To measure microscopic cellular changes, a multiphoton tomography will be used.
  Arms: CO2 laser + HA
Other: Thulium laser + HA — Probands will be treated with a thulium laser. Afterwards a HA gel will be applied. To measure microscopic cellular changes, a multiphoton tomography will be used.
  Arms: Thulium laser + HA

SUMMARY:
* Weakly crossed-linked hyaluronic acid (HA) can be delivered through multiple injections into the dermal and subnormal layer to improve skin quality. However, this treatment comes with multiple bumps for several days.
* Alternatively, HA can be delivered after CO2 laser or thulium laser pretreatment. As microscopic analysis after this treatment is limited, the object of the present study is to investigate the morphological cellular changes after CO2 laser and thulium laser delivered HA into human skin.

ELIGIBILITY:
Inclusion Criteria:

- healthy male and female patients

Exclusion Criteria:

* pregnancy, breast feeding
* open wounds at the area to be treated

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Size of intercellular spaces | 30 minutes and 30 days after treatment.
  Size of intercellular spaces after CO2 or thulium laser treatment compared to control.
Size of keratinocytes | 30 minutes and 30 days after treatment.
  Size of keratinocytes after CO2 or thulium laser treatment compared to control.
Size of hyaluronic acid granules | 30 minutes and 30 days after treatment.
  Size of HA granules after CO2 or thulium laser treatment compared to control.
Distribution of Hyaluronic Acid | 30 minutes and 30 days after treatment.
  Distribution though the epidermal and dermal layers after CO2 or thulium laser treatment compared to control.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical-Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nguyen L, Mess C, Schneider SW, Huck V, Herberger K. In vivo visualisation of tattoo particles using multiphoton tomography and fluorescence lifetime imaging. Exp Dermatol. 2022 Nov;31(11):1712-1719. doi: 10.1111/exd.14646. Epub 2022 Jul 25. PMID 35837813